CLINICAL TRIAL: NCT01602705
Title: Effective Feedback to Improve Primary Care Prescribing Safety (EFIPPS): a Randomised Controlled Trial Using ePrescribing Data
Brief Title: Effective Feedback to Improve Primary Care Prescribing Safety
Acronym: EFIPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); University of Strathclyde (Other); Information Services Division, NHS Scotland (Unknown)
Responsible Party: Principal Investigator, Bruce Guthrie, Professor of Primary Care Medicine, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010PS06
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Complications of Surgical and Medical Care: General Terms
Keywords: Feedback (NOT MESH); Medication errors; Medication review; Inappropriate medication; Randomised controlled trial; Primary Health Care; Family Practice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Placebo Comparator)
  Interventions: Other: Usual care
- Usual care + feedback of practice performance (Active Comparator)
  Interventions: Other: Feedback of Performance
- Usual care + feedback + health psychology intervention (Active Comparator)
  Interventions: Other: Feedback of Performance + Health Psychology Informed Intervention

INTERVENTIONS:
Other: Usual care — Practices in the usual care arm receive a one-off educational newsletter and support for searching for patients in their electronic health record in the form of downloadable searches
  Arms: Usual care
Other: Feedback of Performance — Usual care (educational newsletter and support for searching) plus quarterly feedback of practice rates of high risk prescribing compared to a benchmark of the upper quartile of all practices in the year before
  Arms: Usual care + feedback of practice performance
Other: Feedback of Performance + Health Psychology Informed Intervention — Usual care (educational newsletter + support for searching) plus quarterly feedback plus health psychology informed intervention (persuasive communication and action planning) embedded in feedback
  Arms: Usual care + feedback + health psychology intervention

SUMMARY:
We hypothesise that feedback and feedback + psychology informed intervention delivered to primary care medical practices will reduce high-risk prescribing to patients compared to a simple educational intervention alone. The specific objectives are :

1. To test the effectiveness of the two EFIPPS feedback arms in reducing the specified primary outcome of a composite measure of high-risk antipsychotic, non-steroidal anti-inflammatory drug, and antiplatelet drug prescribing
2. To test the effectiveness of the two EFIPPS feedback arms in reducing the specified secondary outcomes of the six individual measures constituting the composite
3. To assess the cost-effectiveness of the intervention

DETAILED DESCRIPTION:
High risk prescribing is the use of drugs which carry significant risk to patients. Such prescribing is not always inappropriate but does require regular review to ensure that the balance of risk and benefit in individuals is appropriate. High risk prescribing is common and varies widely between practices, and there is evidence that intensive interventions (for example, pharmacist led medication review) can reduce rates of high risk prescribing. The aim of this study is to test whether a simpler and therefore cheaper feedback intervention can reduce high risk prescribing. The study is a three arm cluster randomised trial with primary care medical practices as the unit of randomisation and outcomes measured at patient level using routinely held prescribing for individual patients. The trial will compare two forms of feedback of practice rates of high risk prescribing with usual care. Usual care matches existing NHS working practice. The first active arm will receive quarterly feedback. The second active arm will receive the same feedback plus a health psychology informed intervention designed to promote response to feedback embedded in the feedback.

ELIGIBILITY:
Inclusion Criteria:

* General medical practices in NHS Ayrshire and Arran, NHS Lanarkshire and NHS Lothian

Exclusion Criteria:

* Practices with <250 registered patients
* Practices with <93% of scripts in the new PIS data warehouse having a unique patient identifier (the Community Health Index [CHI] number)
* Practices which were formed after 1st January 2011
* Practices which cease to exist during the trial
* Practices which merge during the trial, where the merging practices were originally in different arms of the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Composite measure of proportion of patients at risk of an adverse event from specified prescribing. | Change in proportion of patients prescribed a high risk drug between baseline and 12 months after the intervention
  The primary outcome is a composite of six high-risk prescribing measures relating to antipsychotic, non-steroidal anti-inflammatory and antiplatelet drug use. It is defined as the proportion of patients particularly at risk of an adverse event from the specified prescribing, who receives one or more high risk prescriptions. A composite is reasonable because each of the underlying indicators is based on evidence of harm and has been judged valid in one or more formal consensus studies, so the composite is a coherent measure of 'high-risk prescribing'.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Guthrie, Principal Investigator — Professor of Primary Care
Locations (1):
- NHS National Services Scotland, Edinburgh, United Kingdom

REFERENCES:
- [Result] Guthrie B, Treweek S, Petrie D, Barnett K, Ritchie LD, Robertson C, Bennie M. Protocol for the Effective Feedback to Improve Primary Care Prescribing Safety (EFIPPS) study: a cluster randomised controlled trial using ePrescribing data. BMJ Open. 2012 Dec 13;2(6):e002359. doi: 10.1136/bmjopen-2012-002359. Print 2012. PMID 23242239
- [Derived] Guthrie B, Kavanagh K, Robertson C, Barnett K, Treweek S, Petrie D, Ritchie L, Bennie M. Data feedback and behavioural change intervention to improve primary care prescribing safety (EFIPPS): multicentre, three arm, cluster randomised controlled trial. BMJ. 2016 Aug 18;354:i4079. doi: 10.1136/bmj.i4079. PMID 27540041
- [Derived] Barnett KN, Bennie M, Treweek S, Robertson C, Petrie DJ, Ritchie LD, Guthrie B. Effective Feedback to Improve Primary Care Prescribing Safety (EFIPPS) a pragmatic three-arm cluster randomised trial: designing the intervention (ClinicalTrials.gov registration NCT01602705). Implement Sci. 2014 Oct 11;9:133. doi: 10.1186/s13012-014-0133-9. PMID 25304255
- See also: Link to open access published protocol — http://bmjopen.bmj.com/content/2/6/e002359.abstract?sid=2efaa72e-9975-448a-b2cf-2ef2c60aff50